CLINICAL TRIAL: NCT00654147
Title: A Pilot Study to Assess Virologic Suppression and Immune Recovery With Raltegravir and Lopinavir/Ritonavir and Raltegravir and Emtricitabine/Tenofovir in HIV-1 Infected Treatment-naïve Subjects
Brief Title: Raltegravir + Lopinavir/Ritonavir or Emtricitabine/Tenofovir for HIV Treatment Naive Subjects
Acronym: HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Margaret A. Fischl, M.D. (Other)
Responsible Party: Sponsor-Investigator, Margaret A. Fischl, M.D., Professor of Medicine, Director AIDS Clinical Research Unit, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A009
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: HIV Infections
Keywords: HIV; antiretroviral therapy naive; Integrase inhibitor; HIV/AIDS; treatment naïve
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium; Lopinavir; Ritonavir; lopinavir-ritonavir drug combination; Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir & Lopinavir/ritonavir (Active Comparator): Raltegravir 400 mg tablet and Lopinavir/ritonavir capsule by mouth, every 12 hours for 48 weeks
  Interventions: Drug: Raltegravir & Lopinavir/ritonavir
- Raltegravir & emtricitabine/tenofovir (Active Comparator): Raltegravir 400 mg tablet bu mouth, every 12 hours for 48 weeks and tenofovir/embritcitabine 200 mg/100 mg table by mouth, once daily for 48 weeks
  Interventions: Drug: Raltegravir and emtricitabine/tenofovir

INTERVENTIONS:
Drug: Raltegravir & Lopinavir/ritonavir — Two drug regimen of an integrase inhibitor and ritonavir boosted protease inhibitor
  Other Names: Isentress; Kaletra
  Arms: Raltegravir & Lopinavir/ritonavir
Drug: Raltegravir and emtricitabine/tenofovir — Three drug regimen of an integrase inhibitor and a fixed dose combination of a non-nucleoside/nucleotide inhibitors
  Other Names: Isentress; Truvada
  Arms: Raltegravir & emtricitabine/tenofovir

SUMMARY:
A prospective, randomized, open-label pilot study to assess virologic suppression and immunologic recovery associated with a two-drug antiretroviral regimen of Raltegravir and the protease inhibitor lopinavir/ritonavir (LPV/r) and a three drug regimen with Raltegravir and two nRTIs (emtricitabine/tenofovir) in HIV-1 infected treatment-naïve subjects.

Immunology Substudy added to determine the kinetics of recovery of CD4 T cells and subpopulations (regulatory T cell [T regs], TH-17 and TH1) after treatment initiation with Raltegravir based regimens and their relationship with functional CD8 T cells and if Raltegravir containing therapies leads to decreases in markers of gut microbial translocation and of cellular and soluble markers of immune activation.

DETAILED DESCRIPTION:
A009 is a prospective, randomized, open-label pilot study to assess virologic suppression and immune recovery rates associated with a two-drug potent antiretroviral regimen of raltegravir and the protease inhibitor lopinavir/ritonavir and a three-drug regimen with raltegravir and two nRTIs (emtricitabine/tenofovir) in treatment-naïve subjects.

HIV-1-infected subjects who are antiretroviral drug-naïve and have plasma HIV-1 RNA levels ≥5000 copies/ml obtained within 30 days prior to study entry will be randomized 1:1 to Raltegravir 400 mg BID + LPV 400 mg/RTV 100 mg BID (Arm A) or Raltegravir 400 mg BID + FTC 200 mg/TDF 300 mg QD (Arm B).

Subjects will have measurements of HIV-1 RNA and CD4+ and CD8+ T-cell counts at pre-entry and entry. The average of these measurements will be used to establish their baseline values. Following entry, subjects will have plasma HIV-1 RNA samples drawn at days 2, 4, 8 and at weeks 2, 4, 8, 16, 24, 32, 40 and 48 and at virologic failure. CD38 expression on CD4+/CD8+ cells and CD38/HLA-DR activation antigen on CD4+ and CD8+ cells and subsets T-cell percentage will be done at entry, day 8 and weeks 4, 8, 24 and at virologic failure by advanced flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV Infection
* Genotypic resistance without major resistance mutations within 30 days
* Antiretroviral drug-naïve
* Screening HIV-1 RNA ≥5000
* Women of reproductive potential
* Negative pregnancy test within 48 hours

Exclusion Criteria:

* Acute or recent HIV-1 infection
* Currently breast feeding
* Use of immunomodulators
* Evidence of major resistance mutations
* HBsAg positive
* Acute hepatitis of any etiology or clinically significant liver disease
* Current imprisonment or involuntary incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A Fischl, M.D., Study Chair — University of Miami AIDS Clinical Research Unit
Locations (1):
- University of Miami AIDS Clinical Research Unit, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomly assigned to receive one of two regimens Raltegravir (Isentress, Merck & Company) 400 mg twice daily with either Lopinavir/ritonavir (Kaletra, Abbott Laboratories) 200 mg/100 mg twice daily or with emtricitabine/tenofovir (Truvada, Gilead Sciences) 200 mg/100 mg twice daily.
Pre-assignment Details: Participants with acute or recent HIV-1 infection, major resistance-associated mutation on any genotype performed at any time prior to study entry, serious illness requiring systemic treatment and/or hospitalization within 7 days of study entry, HBsAg positivity, acute hepatitis of any etiology, clinically significant liver disease were excluded
Groups:
- Raltegravir & Lopinavir/Ritonavir: Raltegravir 400 mg tablet and Lopinavir/ritonavir 400 mg/100 mg capsules every 12 hours for 48 weeks
  Raltegravir and Lopinavir/ritonavir: 400 mg BID for 48 weeks 400mg/100 mg BID for 48 weeks
- Raltegravir & Emtricitabine/Tenofovir: Raltegravir 400 mg tablet every 12 hours & emtricitabine 200mg/tenofovir 300 mg tab once daily for 48 weeks
  Raltegravir, emtricitabine, tenofovir: 400 mg BID for 48 weeks 200 mg QD for 48 weeks 300 mg QD for 48
Period: Overall Study
Arm/Group | Raltegravir & Lopinavir/Ritonavir | Raltegravir & Emtricitabine/Tenofovir
Started | 21 | 23
Completed | 19 | 19
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Raltegravir & Lopinavir/Ritonavir: Raltegravir 400 mg tablet every 12 hours for 48 & Lopinavir/ritonavir 400 mg/100 mg capsules every 12 hours for 48 weeks
  Raltegravir and Lopinavir/ritonavir: 400 mg BID for 48 weeks 400mg/100 mg BID for 48 weeks
- Raltegravir & Emtricitabine/Tenofovir: Raltegravir 400 mg tablet every 12 hours for 48 weeks & emtricitabine 200mg/ tenofovir 300 mg tab once daily for 48 weeks
  Raltegravir, emtricitabine, tenofovir: 400 mg BID for 48 weeks 200 mg QD for 48 weeks 300 mg QD for 48
- Total: Total of all reporting groups
Arm/Group | Raltegravir & Lopinavir/Ritonavir | Raltegravir & Emtricitabine/Tenofovir | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 23 | 44
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 18 | 22 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 15 | 28
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 12 | 16 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Time to Confirmed Virologic Failure
Description: time to confirmed viologic failure at 24 weeks (up to 48 weeks)
Time Frame: weeks
Population: descriptive
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Raltegravir & Lopinavir/Ritonavir | Raltegravir & Emtricitabine/Tenofovir
Number analyzed (Participants) | 21 | 23
weeks | 28 [25 to 56] | 29 [21 to 56]

2. Secondary Outcome: Study Medication Toxicity-related Discontinuation .
Description: grade 3 and grade 4 symptoms and laboratory study treatment limiting toxicity
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | Raltegravir & Lopinavir/Ritonavir | Raltegravir & Emtricitabine/Tenofovir
Number analyzed (Participants) | 21 | 23
participants | 1 | 0

3. Secondary Outcome: Weeks to HIV-1 RNA <200 Copies/ml
Description: time to viral suppression noted as week on study treatment to attain HIV-1 RNA < 200 copies/ml
Time Frame: from date of treatment start to first week documented viral suppression
Measure: Median (95% Confidence Interval); unit: week to viral supresssion
Arm/Group | Raltegravir & Lopinavir/Ritonavir | Raltegravir & Emtricitabine/Tenofovir
Number analyzed (Participants) | 21 | 23
week to viral supresssion
  week to <200 Copies/ml | 28 [14 to 56] | 28 [14 to 33]
  week to <50 Copies/ml | 56 [28 to 108] | 56 [28 to 57]

4. Secondary Outcome: Change From Baseline CD4+ and CD8+ Cell Counts
Description: mean change in CD4+ and CD8+ T-lymphocytes counts from baseline (defined as the average of pre-entry and entry values) at weeks 16 and 24 in the two treatment arms
Time Frame: Baseline, Weeks 16 and 24
Population: Change from baseline compared between arms using repeated measures analysis of covariance. Linear mixed models used to accomplish these analyses.
Measure: Mean (Standard Error); unit: cells/mm3
Arm/Group | Raltegravir & Lopinavir/Ritonavir | Raltegravir & Emtricitabine/Tenofovir
Number analyzed (Participants) | 21 | 23
cells/mm3
  week 16 CD4 cells | 516.34 (76.52) | 452.11 (92.48)
  week 24 CD4 cells | 521.31 (76.52) | 482.36 (93.32)

5. Secondary Outcome: Study Medication Tolerability
Description: study treatment tolerability as measured by number of subjects receiving study treatment who either discontinued or changed any component of study treatment
Time Frame: date started study treatment to first week documented change study treatment up to week 48
Measure: Number; unit: participants
Arm/Group | Raltegravir & Lopinavir/Ritonavir | Raltegravir & Emtricitabine/Tenofovir
Number analyzed (Participants) | 21 | 23
participants | 1 | 0

6. Primary Outcome: Time to Virologic Failure
Description: time to virologic failure at week 24 (up to 48 weeks)
Time Frame: week 24 (up to 48 weeks)
Measure: Median (Standard Deviation); unit: weeks
Arm/Group | Raltegravir & Lopinavir/Ritonavir | Raltegravir & Emtricitabine/Tenofovir
Number analyzed (Participants) | 21 | 23
weeks | 3.2296 (0.1596) | 2.9952 (0.1812)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Raltegravir & Lopinavir/Ritonavir | Raltegravir & Emtricitabine/Tenofovir
Serious Adverse Events (participants affected / at risk) | 4/21 | 0/23
Other Adverse Events (participants affected / at risk) | 1/21 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir & Lopinavir/Ritonavir (N=21) | Raltegravir & Emtricitabine/Tenofovir (N=23)
Total bilirubin (Hepatobiliary disorders) | 2 (2) | 0 (0) — grade 3 or greater elevation in total bilirubin
trigylcerides (Endocrine disorders) | 2 (3) | 0 (0) — grade 3 or greater elevation in fasting blood triglycerides
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir & Lopinavir/Ritonavir (N=21) | Raltegravir & Emtricitabine/Tenofovir (N=23)
nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Pilot study with 44 subjects and generalization f results is limited by the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No